CLINICAL TRIAL: NCT03783741
Title: The Biopsychosocial Burden of Prostate Biopsy at the Time of Its Indication, Procedure, and Pathological Report
Brief Title: The Biopsychosocial Burden of Prostate Biopsy
Status: Completed | Type: Observational
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Leonardo Oliveira Reis, Professor, University of Campinas, Brazil
Other Study IDs: Prostate Biopsy Burden
Record Dates: First submitted 2018-12-17; First posted 2018-12-21 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Biopsy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Questionnaire — Interview

SUMMARY:
Prostate biopsy was offered to 47 consecutive patients with prostate-specific antigen (PSA) over 4 ng/dl or suspicious digital rectal examination (DRE) of whom 16 had undergone a biopsy. Comprehensive validated questionnaires at TIME 0 (pre-biopsy), TIME 1 (before diagnosis, 20 days after biopsy) and TIME 2 (after diagnosis, 40 days after biopsy) accessed patients' erectile (IIEF-5) and voiding (IPSS) functions, Beck scales measured anxiety (BAI), hopelessness (BHS) and depression (BDI), added to the emotional thermometers including five visual analog scales for distress, anxiety, depression, anger and need for help. Mann-Whitney or Friedman tests were obtained among times and studied variables.

DETAILED DESCRIPTION:
A prospective, longitudinal and observational study in which the sexually active patients were evaluated in the Urology Department of the city of Paulínia, submitted to biopsy guided by transrectal ultrasound after ethics committee approval (355.357).

Consecutive patients who were attended by urologist and present prostate cancer suspicions (PSA> 4 ng / dL and/or rectal examination (TR) were submitted a BXP. They were evaluated at three different moments of the biopsy:

* Seven days before the biopsy procedure (T0);
* 20 days after the biopsy, upon receiving the histopathological result, before becoming aware of it (T1);
* 40 days after the biopsy, 20 days after being aware of the test result (T2). Sixty-one consecutive patients were invited to participate in the study, 10 of them had no active sexual life and 9 answered the questionnaires only at the first moment, were excluded; 47 responded at three times (T0, T1, and T2).

Validated instruments were applied - IIEF-5 (erectile function); - IPSS (voiding function); - Beck scales - BAI (anxiety), BHS (hopelessness), BDI (depression); and - Emotional thermometers.

The comparison among the moments (T0, T1, and T2) was performed through Friedman (analysis of variance) for repeated measures with the variables transformed in stations. The comparison between patients and variables was performed using the Mann-Whitney test. The sample power was calculated and the level of significance considered was 5%.

ELIGIBILITY:
Inclusion Criteria:

* prostate cancer suspicion (PSA > 4 ng / dL, digital rectal examination)

Exclusion Criteria:

* not agree to participate

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Consecutive patients who were attended by a urologist with prostate biopsy indication.
Sampling Method: Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Erectile Function | Change from time of biopsy indication (T0) compared to 20 days after procedure (T1) and 20 days after pathological report result (T2, 40 days)
  International Index of Erectile Function - IIEF-5 index (range 0-25; higher better)
Voiding Function | Change from time of biopsy indication (T0) compared to 20 days after procedure (T1) and 20 days after pathological report result (T2, 40 days)
  International Prostatic Symptoms Score - IPSS (range 0-35; higher worse)
Beck scale | Change from time of biopsy indication (T0) compared to 20 days after procedure (T1) and 20 days after pathological report result (T2, 40 days)
  Beck Anxiety Index - BAI (0-63; higher worse)
Emotional thermometers | Change from time of biopsy indication (T0) compared to 20 days after procedure (T1) and 20 days after pathological report result (T2, 40 days)
  Thermometer score (range 0-10; higher worse)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas Unicamp, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Naccarato AM, Reis LO, Matheus WE, Ferreira U, Denardi F. Barriers to prostate cancer screening: psychological aspects and descriptive variables---is there a correlation? Aging Male. 2011 Mar;14(1):66-71. doi: 10.3109/13685538.2010.522277. Epub 2010 Oct 12. PMID 20937009
- [Derived] Laranja WW, Sanches BCF, Voris BRI, Alonso JCC, Simoes FA, Rejowski RF, Reis LO. The Biopsychosocial Burden of Prostate Biopsy at the Time of Its Indication, Procedure, and Pathological Report. Prostate Cancer. 2019 Apr 1;2019:2653708. doi: 10.1155/2019/2653708. eCollection 2019. PMID 31057971